CLINICAL TRIAL: NCT00027989
Title: An Open-Label, Single-Arm, Phase II Study of Liposomal Doxorubicin (Doxil) and Gemcitabine in the Treatment of Women With Metastatic Breast Cancer
Brief Title: Liposomal Doxorubicin and Gemcitabine in Treating Women With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pharmatech Oncology (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069104; PHARMATECH-P01-00002008; ORTHO-PHARMATECH-P01-000020008; PHARMATECH-20002183
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2004-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of combining liposomal doxorubicin with gemcitabine in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in women with metastatic breast cancer treated with doxorubicin HCl liposome and gemcitabine.
* Determine the duration of response, time to disease progression, and duration of survival of patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the quantitative toxicity of this regimen, in terms of incidence, type, and severity, in these patients.

OUTLINE: This is a multicenter study.

Patients receive doxorubicin HCl liposome IV over 1 hour on day 1 and gemcitabine IV over 30 minutes on days 1 and 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 2 courses beyond documentation of CR.

Quality of life is assessed at baseline, on day 1 of each course, and then at the end of study.

Patients are followed at 4 weeks and then every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic breast cancer
* Measurable disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL
* Absolute neutrophil count at least 1,500/mm^3
* No impaired bone marrow function

Hepatic:

* Bilirubin no greater than 2 mg/dL
* AST and ALT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN (unless attributed to tumor)
* No impaired hepatic function

Renal:

* Creatinine no greater than 2.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No impaired renal function

Cardiovascular:

* No prior cardiac disease within the past 5 years OR
* LVEF at least 50%

Other:

* No prior uncontrolled seizures
* No uncontrolled systemic infection
* No anthracycline resistance
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior trastuzumab (Herceptin)

Chemotherapy:

* Prior adjuvant therapy with anthracycline of no more than 320 mg/m^2 allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to more than 1/3 of hematopoietic sites

Surgery:

* Not specified

Other:

* At least 30 days since prior investigational medications and recovered
* No more than 1 prior treatment regimen for metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Marcus, Study Chair — Pharmatech Oncology
Locations (5):
- United States (5):
  - Montgomery Cancer Center, Montgomery, Alabama
  - California Cancer Medical Center, West Covina, California
  - Pharmatech Oncology, Denver, Colorado
  - Oncology-Hematology Associates, P.A., Clinton, Maryland
  - South Carolina Oncology Associates, Columbia, South Carolina